CLINICAL TRIAL: NCT03894436
Title: Ultrasound-Guided Diaphragmatic Thickness Assessment as an Indicator of Successful Extubation in Mechanically Ventilated Cancer Patients
Brief Title: Ultrasound-Guided Diaphragmatic Thickness Assessment as an Indicator of Successful Extubation in Mechanically Ventilated
Status: Completed | Type: Observational
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Soliman, Assestant lecturer of anaesthesia,icu and pain management, National Cancer Institute, Egypt
Other Study IDs: IRB00004025
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Successful Weaning; Weaning Failure
MeSH Terms: interventions — Blood Gas Analysis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: Ultrasound assessment of diaphragm thickness in B-mode — assess the thickness of diaphragm needed as a tool for prediction of extubation and proper timing of weaning from mechanical ventilation in the ICU which is measured by B mode ultrasound in ventilated cancer patients
  Other Names: Rapid shallow breathing index; Arterial blood gases

SUMMARY:
Weaning of mechanically ventilated patient is a daily challenge in Intensive Care units. Several indexes have been employed to assess the patient's ability to recover efficient spontaneous breathing. As the diaphragm is the main respiratory muscle, direct measurement of diaphragmatic function as predictors of extubation success or failure have not been extensively evaluated. Ultrasound can easily access diaphragm thickness (tdi) in its zone of apposition during, tdi can represent the contractile activity of the diaphragm and the efficiency of its function.

DETAILED DESCRIPTION:
Each patient will have an orotracheal tube, and will be mechanically ventilated in pressure support ventilation (PSV) mode according to the clinical needs. Local guidelines for sedation of postoperative patients prescribe the use of an intravenous (iv) continuous infusion of propofol, starting at 1.5 mg/kg/h and titrated to obtain a Richmond agitation-sedation scale (RASS) score of 0/-1. Analgesia is provided as a 6- to 8-ml/h continuous epidural infusion of bupivacaine 0.125% + fentanyl 2-mcg/ml solution, aiming at a verbal numerical rating <4 or a behavioral pain scale <7. If epidural analgesia is not feasible, patients receive 0.5 to 1 mg/kg/h continuous iv infusion of morphine + iv acetaminophen 1 g three/four times per day. Patients enrolled when judged to be eligible for a test of weaning from mechanical ventilation, following the local weaning guidelines, that is, adequate cough, absence of excessive tracheobronchial secretion, clinical stability, heart rate (HR) <140/min, systolic blood pressure between 90 and 140 mmHg, arterial partial pressure of oxygen/inspired oxygen fraction (PaO2/FIO2) ≥150 mmHg, respiratory rate <35/min, maximal inspiratory pressure < -20 cmH2O, respiratory rate/tidal volume ratio <105 breaths/(min/l) [19]. Weaning trials consisted of spontaneous breathing(SB) trials on PS mode (reducing PS by 5 cm H2O until a PS level of Δ5/5 was obtained). A successful extubation will be defined as SB for >48 h following extubation. A failed extubation will be defined as reintubation within 48 h. The RSBI (f in breaths/minute (f)/tidal volume in liters (VT)will be calculated simultaneously with ultrasound measurements of tdi and simultaneously with other criteria for weaning.

TECHNIQUE Diaphragm thickness (tdi) was measured using a 6-13 MHz linear ultrasound probe set to B mode (SonoSite M-turbo ultrasound machine). The right hemidiaphragm was imaged at the zone of apposition of the diaphragm and rib cage in the midaxillary line between the 8th and 10th intercostal spaces as previously described.[18] All patients were studied with the head of bed elevated between 20° and 40°. The tdi was measured at end-expiration and end-inspiration. The percent change in tdi between end-expiration and end-inspiration (Δtdi%) was calculated as (tdi end-inspiration-tdi end-expiration/tdi end-expiration) ×100. The Δtdi% for each patient represented the mean of three to five breaths. Images were obtained within the first 5 min of the PS trial and immediate before extubation. Data will be collected: 1. Diaphragmatic thickness. 2. The percent change in tdi between end-expiration and end-inspiration Δtdi%. 3. Arterial blood gases (ABG). 4. Rapid Shallow Breathing Index (RSBI) = Respiratory rate/Tidal volume. 5. Duration of ventilator treatment. 6. Success and failure rate of weaning. 7. Body mass index (BMI).

ELIGIBILITY:
Inclusion Criteria:

* Age18-65 years.
* ASA class 1 to 3,
* body mass index (BMI) between 20 and 40 kg/m2
* intubation for ≥ 48 hours
* Types of abdominal cancer surgery included partial gastrectomy, hysterectomy, Splenectomy, hepatectomy, and colectomy.

Exclusion Criteria:

* Hemodynamic instability requiring vasopressors.
* Gas exchange impairment requiring positive end-expiratory pressure (PEEP) >10 cmH2O and/or FIO2 > 50% to obtain a PaO2 > 60 mmHg.
* Pressure support (PS) level > 20 cmH2O.
* Body temperature > 38°C or < 35°C.
* Deep sedation state (RASS score < -1).
* History of chronic obstructive pulmonary disease, neuromuscular disease, anatomical malformation of the diaphragm, or use of muscle paralyzing agents, aminoglycosides and corticosteroids.
* Pneumothorax or pneumomediastinum, increase intrabdominal pressure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fifty patients were recruited during the immediate postoperative period after major elective cancer surgery who needed mechanical ventilation (MV) due to a respiratory cause and met criteria for a spontaneous breathing trial with pressure support ventilation and diaphragm thickness is assessed by using b-mode ultrasound.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2018-08-25 (Actual); Study Completion 2018-11-21 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of diaphragm thickness compared to ABG as standard for weaning | 6 months
  diagnostic accuracy of diaphragm thickness to predict weaning compared to ABG
Sensitivity and specificity of diaphragm delta tdi compared to ABG as standard for weaning | 6 months
  diagnostic accuracy of diaphragm delta tdi to predict weaning compared to ABG

SECONDARY OUTCOMES:
Sensitivity and specificity of RSBI compared to ABG as gold standard for weaning | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Mohamed Soliman, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided